CLINICAL TRIAL: NCT00554411
Title: Assessing Changes at the Ocular Surface Following the Switch From Xalatan to Travatan Z.
Brief Title: Assessing Ocular Surface Changes After Changing Glaucoma Medications
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 07-0757
Record Dates: First submitted 2007-11-02; First posted 2007-11-06 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Glaucoma; Monotherapy With Xalatan From 1 to 18 Months; Ocular Surface Disease
Keywords: Travatan Z; glaucoma; tear film break up time
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Hypothesis: Changing to Travatan Z therapy increases the tear film break up time of subjects on Xalatan therapy presenting with ocular surface disease.

DETAILED DESCRIPTION:
Patients who have been taking Xalatan monotherapy to treat their glaucoma and presenting with ocular surface disease will be advised to switch their medication to Travatan Z. Test results will be recorded at the day that the medication was changed and at follow-up to determine if there is a measurable change in tear film break up, corneal staining and in the Ocular Surface Disease Index.

ELIGIBILITY:
Inclusion Criteria:

* on Xalatan monotherapy from 1 to 18 months
* 18 years of age or older
* has been diagnosed with ocular surface disease

Exclusion Criteria:

* special populations such as children, pregnant females, prisoners, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients will be selected from the ophthalmology clinic of the principal investigator
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2007-11; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Change in Signs and Symptoms of Ocular Surface Disease | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Malik Y Kahook, M.D., Principal Investigator — Rocky mountain Lions Eye Institute
Locations (1):
- Rocky Mountain Lions Eye Institute, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No